CLINICAL TRIAL: NCT02027506
Title: DIAGNOSTIC VALUE OF ELECTROCARDIOGRAPHIC ST-T WAVE CHANGES IN LEAD aVL IN PATIENTS WITH CHRONIC STABLE ANGINA
Brief Title: Diagnostic Value of Electrocardiographic St-t Wave Changes in Patients With Chronic Stable Angina
Acronym: ECG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Awad Youssef Awad Zeid, M.B,CH.B., Alexandria University
Other Study IDs: dvavl2185
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Ekg Change Ischemia Lateral
Keywords: ECG; aVL; CHRONIC STABLE ANGINA; T WAVE
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The electrocardiogram (ECG) is a simple and non-invasive bedside diagnostic tool with a well-established role in the diagnosis of (CAD). Many studies have found that the admission of ECG provides important prognostic information in patients admitted with chest pain. For instance, T wave inversion in anterior or inferior location and or ST-segment depression has been associated with high incidence of CAD.

DETAILED DESCRIPTION:
The aim of the work will be directed to study the diagnostic value of electrocardiographic ST-T wave changes in lead aVL in patients with chronic stable angina

The ECG findings vary considerably, depending importantly on four major factors: (1) the duration of the ischemic process (acute versus evolving or chronic) ; (2) its extent (large versus small) ; (3) its topography (anterior versus inferior-posterior and right ventricular) ; (4) the presence of other underlying conditions (e.g. LBBB, WPW or pacemaker pattern) that can mask or alters the classic pattern.

The resting electrocardiogram is normal in approximately half of patients with chronic stable angina pectoris, and even patients with severe CAD may have a normal tracing at rest. A normal resting ECG suggesting a normal LV function and it is unusual finding in a patient with an extensive previous infarction.

The most common electrocardiographic abnormalities in patients with chronic CAD are non specific ST-Twave changes with or without abnormal Q waves. In addition to myocardial ischemia, other conditions that can produce ST-T wave abnormalities include LV hypertrophy or dilation, electrolyte abnormalities, neurogenic effects, and anti-arrhythmic drugs.

In patients with known CAD, however, the occurrence of ST-T wave abnormalities on the resting ECG may correlate with the severity of the underlying heart disease. This association may explain the adverse association of ST-Twave changes with prognosis of these patients. In contrast, a normal resting ECG is more favorable long-term prognostic sign in patients with suspected or definite CAD.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted at the Alexandria university hospitals or referred from secondary hospitals with documented CAD as proved by non invasive tests

Exclusion Criteria:

* Clinical situations that may result in secondary aVL lead T wave inversion and /or ST segment depression from analysis as Bundle branch block either left or right, aortic stenosis, left ventricular hypertrophy and strain and paced ventricular rhythms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a prospective observational study conducted on 150 patients admitted at the Alexandria university hospitals or referred from secondary hospitals with documented CAD as proved by non invasive tests (ECG, echocardiography, treadmill exercise, myocardial perfusion imaging or multi-slice CT coronary angiography) requiring invasive coronary angiography.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-10 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Corelation between ecg finding and coronary angiography finding | 9 months
  the value of t wave and st segment changes in correlation with the cornary angiographic findings

CONTACTS AND LOCATIONS:
Overall Officials: A Y zeid, M.B,CH.B., Principal Investigator — Alexandria University
Locations (1):
- Alexandria Medical College, Alexandria, Egypt